CLINICAL TRIAL: NCT06305949
Title: A Multi-center, Randomized, Double-blind, Pilot Study to Evaluate the Safety and Efficacy of Optimized Transcranial Direct Current Stimulation for the Transitory Improvement of Swallowing Function in Patients With Post-stroke Dysphagia
Brief Title: Clinical Trial on the Safety and Efficacy of Optimized Transcranial Direct Current Stimulation for the Swallowing Function in Patients With Post-Stroke Dysphagia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NEUROPHET (Industry)
Collaborators: Bucheon St. Mary's Hospital (Other); Saint Vincent's Hospital, Korea (Other); National Traffic Injury Rehabilitation Hospital (Unknown); Pusan National University Yangsan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XC23DDDS0098
Record Dates: First submitted 2024-02-26; First posted 2024-03-12 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-05

CONDITIONS: Deglutition Disorders
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimized transcranial Direct Current Stimulation (Experimental): Patients receive optimized stimulation obtained from an individualized T1 MRI-based simulation of transcranial direct current stimulation for 30 minutes, once a day for 4 weeks, for a total of 20 sessions.
  Interventions: Device: Optimized transcranial Direct Current Stimulation
- Sham transcranial Direct Current Stimulation (Sham Comparator): Patients receive sham stimulation for 30 minutes, once a day for 4 weeks, for a total of 20 sessions.
  Interventions: Device: Sham transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Optimized transcranial Direct Current Stimulation — transcranial Direct Current Stimulation 2mA for 30 min; The anode electrode will be located over the contralesional representation of the motor cortex swallowing area, while the cathode electrode will be positioned on the ipsilesional side
  Other Names: NEUROPHET tES LAB; NEUROPHET innk01-DW
  Arms: Optimized transcranial Direct Current Stimulation
Device: Sham transcranial Direct Current Stimulation — transcranial Direct Current sham Stimulation for 30 min; The anode electrode will be located over the contralesional representation of the motor cortex swallowing area, while the cathode electrode will be positioned on the ipsilesional side
  Other Names: NEUROPHET tES LAB; NEUROPHET innk01-DW
  Arms: Sham transcranial Direct Current Stimulation

SUMMARY:
The goal of this clinical trial is to evaluate whether the application of optimized transcranial direct current stimulation is more effective compared to sham stimulation for temporary improvement of swallowing function in patients with post-stroke dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* men and women >19 years old
* patients with stroke confirmed by neuroimaging
* first-time stroke patients
* patients in subacute or chronic phases of stroke with 3 weeks or more after onset
* stroke patients with confirmed dysphagia through Videofluoroscopic Swallowing Study (VFSS).

Exclusion Criteria:

* patients with recurrent stoke, traumatic brain injury, spine cord injury, and degenerative brain disease, such as Parkinson's disease, etc.
* patients with deteriorated cognitive function unable to perform the clinical trial as instructed
* patients with evidence of delirium, confusion, or other impairment of consciousness
* patients with uncontrolled medical disease or surgical conditions
* patients ineligible for Transcranial direct current stimulation (due to scalp condition, metallic material at the electrode attachment area, presence of a pacemaker or cochlear implant)
* patients with previous experience within the last year using a stimulation device similar to the one use in this clinical trial or who have participated in related clinical trials
* patients with severe neurologic disorder with concomitant major psychiatric disorder such as major depressive disorder and dementia
* patients with history of uncontrolled epilepsy within 6 months
* patients with medical contraindications for neuroimaging test, such as MRI;
* patients who are taken contraindicated medications or require medication changes during the trial period that could influence cognitive/motor function changes via brain activation changes
* patients who are pregnant, breastfeeding, or planning pregnancy during the trial period
* patients considered medically ineligible for participation in the present trial beyond the criteria listened above.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Functional Oral Intake Scale (FOIS) | Baseline, At 4 weeks from baseline
  FOIS is a scale used for purposes to assess changes in functional oral intake of food and liquids in patients with dysphagia. FOIS is sensitive to changes in oral intake of food and liquid over time in stroke patients. The scale ranges from level 1 (nothing by mouth) to level 7 (a full unrestricted oral diet)
Penetration-aspiration Scale (PAS) | Baseline, At 4 weeks from baseline
  PAS is a standard scale to assess deglutition in clinical practice and research. It is composed of an 8-point scale used to characterize both the location of airway invasion events and patient's response during video fluoroscopic swallowing studies. The scale design to capture three constructs: depth of airway invasion, material remaining after swallow, and patient's response to aspiration. The scale ranges from score 1 (Material does not enter the airway) to score 8 (Material enters the airway, passes below the level of the vocal folds, and no effort is made to eject)

SECONDARY OUTCOMES:
Functional Oral Intake Scale (FOIS) | Baseline, At 2, 4, and 8 weeks from baseline
  FOIS is a scale used for purposes to assess changes in functional oral intake of food and liquids in patients with dysphagia. FOIS is sensitive to changes in oral intake of food and liquid over time in stroke patients. The scale ranges from level 1 (nothing by mouth) to level 7 (a full unrestricted oral diet)
Penetration-aspiration Scale (PAS) | Baseline, At 2, 4, and 8 weeks from baseline
  PAS is a standard scale to assess deglutition in clinical practice and research. It is composed of an 8-point scale used to characterize both the location of airway invasion events and patient's response during video fluoroscopic swallowing studies. The scale design to capture three constructs: depth of airway invasion, material remaining after swallow, and patient's response to aspiration. The scale ranges from score 1 (Material does not enter the airway) to score 8 (Material enters the airway, passes below the level of the vocal folds, and no effort is made to eject)
Videofluoroscopic Dysphagia Scale (VDS) | Baseline, At 2, 4, and 8 weeks from baseline
  The scale contains 14 categories that represent both oral functions (lip, closure, mastication , bolus formation, premature bolus loss, apraxia and oral transit time) and pharyngeal functions (pharyngeal triggering, laryngeal elevation, epiglottic closure, pharyngeal transit time, pharyngeal coating, vallecular and pyriform sinus residues, and tracheal aspiration), with a sum of 100 points.
Korean Mann Assessment of Swallowing Ability (K-MASA) | Baseline, At 2, 4, and 8 weeks from baseline
  K-MASA assesses 24 skills related to sensory and oral motor elements of swallowing. Performance for each skill is measured using a 5- or 10-points rating scale and tallied to create a total numeric score out of 200 possible points, which are interpreted as no abnormality (≥178), mild dysphagia (168-177), moderate dysphagia (139-167) and severe (≤138)
Speech Mechanism Screening Test (SMST) | Baseline, At 4, and 8 weeks from baseline
  The test consists of 13 questions to evaluate the structure of the articulatory system, including the face, lips, tongue, jaw, teeth, oral cavity, soft palate, pharynx, and breathing; 17 questions to evaluate the function of the articulatory system; 3 questions to auditorily evaluate the structure and function of the vocal system; and 14 questions to evaluate the regularity and articulation accuracy of the mutual movement of the articulatory system during articulatory alternation.
Urimal Test of Articulation and Phonology (U-TAP) | Baseline, At 4, and 8 weeks from baseline
  U-TAP is a test designed for native speakers of the Korean language. It is aimed to evaluate the pronunciation produced in words and sentences by patients with speech sound disorders who have problems with consonant or vowel sounds. It is recorded by phonological word and syllable position and calculates consonant accuracy and word-level phonological indices at the word and sentence levels to compare with normal articulation development
modified Rankin Scale (mRS) | Baseline, At 2, 4, and 8 weeks from baseline
  mRS is composed of a 6-point assessment that includes reference to both limitations in activity and changes in lifestyle. The mRS possible scores vary from 0 (no symptoms) to 6 (dead) points
Gugging Swallowing Screen | Baseline, At 2, 4, and 8 weeks from baseline
  The assessment is composed of two parts, the preliminary assessment (indirect swallowing test) and the direct swallowing test, which consist of 4 items with 3 subtests (semisolid, liquid and solid). The test is based on a pointing system where higher numbers denote better performance, with a maximum of 5 points that can be reached in each subtest.
Eating Assessment Tool-10 (EAT-10) | Baseline, At 2, 4, and 8 weeks from baseline
  The EAT-10 is a tool to assess self-perceived symptoms of oropharyngeal dysphagia and monitor changes in response to a treatment. It consists of ten items to be rated on a 5-point response scale (0-4), with "0" = No problem and "4" = Severe problem, the maximum score possible is 40.
Iowa Oral Performance Instrument (IOPI) | Baseline, At 4, and 8 weeks from baseline
  IOPI is a standardized portable device that is used to quantify tongue and lips isometric strength and endurance.
Motor-Evoked Potential (MEP) | Baseline, At 2 and 4 weeks from baseline
  The cortical excitability of the area corresponding to the swallowing movement will be assessed by changes in the amplitude and latency of the MEPs by using transcranial magnetic stimulation (TMS).
Grade, Roughness, Breathiness, Asthenia and Strain scale(GRBAS scale) | Baseline, At 4, and 8 weeks from baseline
  GRBAS scale is used by researchers and clinicians for rating voice quality using a 4-point Likert scale with the following judgments: 0 = normal, 1 = mild impairment, 2 = moderate impairment, and 3 = severe impairment.
Respiratory muscle strength | Baseline, At 4, and 8 weeks from baseline
  Respiratory muscle strength will be assessed by maximal inspiratory and expiratory pressure
Peak cough flow | Baseline, At 4, and 8 weeks from baseline
  Peak cough flow measures the maximum expiratory flow during the compressive phase of a cough just after sudden opening of the glottis

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea, Bucheon St. Mary's Hospital, Bucheon-si, South Korea